CLINICAL TRIAL: NCT04306809
Title: Internet-delivered ACT for PTSD and Chronic Pain : a Development Pilot Series
Brief Title: iACT for PTSD and Chronic Pain : a Development Pilot Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Sophia Åkerblom, Prinicpal Investigator, Skane University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SkaneU2020
Record Dates: First submitted 2020-02-20; First posted 2020-03-13 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2021-10

CONDITIONS: PTSD; Chronic Pain
Keywords: PTSD; Chronic pain
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Internet delivered Acceptance and Commitment Therapy for PTSD and Chronic Pain, supported by a psychologist
  Interventions: Behavioral: Internet-delivered ACT for PTSD and chronic pain

INTERVENTIONS:
Behavioral: Internet-delivered ACT for PTSD and chronic pain — The participants will go through an active internet-based ACT treatment focused on education about PTSD, value-based exposure for the traumatic memory and avoided situations, and behavior change through exercises targeting the processes mindfulness, cognitive defusion and acceptance. The treatment is delivered on a safe internet platform. Participants have planned telephone contact with their assigned psychologist 3 times during the program and can also contact their psychologist via a message system in the platform and expect answer within 48 hours.

SUMMARY:
The primary aim of this study is to investigate the effect of Internet-delivered Acceptance and commitment therapy for PTSD and comorbid chronic pain. First, a pilot study (no randomization; N=10) will be conducted to test the intervention and assessment procedures. This will be followed by a randomized controlled trial with waitlist control. The participants will go through an active internet-based ACT treatment focused on education about PTSD, value-based exposure for the traumatic memory and avoided situations, and behavior change through exercises targeting the processes mindfulness, cognitive defusion and acceptance. The treatment is delivered on a safe internet platform. Participants have planned telephone contact with their assigned psychologist 3 times during the program and can also contact their psychologist via a message system in the platform and expect answer within 48 hours.

DETAILED DESCRIPTION:
Objective: The primary aim of this study is to investigate the effect of Internet-delivered Acceptance and commitment therapy (iACT) for PTSD and comorbid chronic pain.

Sample size: 10 participants.

Trial design: All participants are offered treatment. Participants are recruited from the Pain Rehabilitation Unit at Skåne University Hospital. The unit is a government supported, regional specialist center focused on assessment and treatment of chronic pain and related disability.

Assessments: Baseline and post treatment (2 weeks after treatment) assessments will be conducted by an assessor who is trained to administer the study measures. Self-report measures will also collected at this time, post treatment (2 weeks after treatment) as well as during a 3-month follow up.

Assessment includes:

Pre-and post assessment: Assessors will collect demographic information, self-report measures, and trauma history. During the pre- and post-assessment the Clinician-Administered PTSD Scale for DSM-5 will be administered to establish PTSD whether participants met the DSM-5 criteria for PTSD.

During the pre-assessment the Mini International Neuropsychiatric Interview 5.0 (MINI) will be administered to detect the presence of other comorbid disorders and assess inclusion criteria and rule out exclusion criteria.

Post-treatment exit interview: At the post-assessment, the assigned assessor will ask participants about their satisfaction with and experience of the program, what they found helpful or unhelpful and suggestions for future improvements.

During treatment: During treatment the treatment credibility scale will be administered to assess the patients' perceptions of how credible the treatment is following the introduction of the treatment rationale and the main treatment components (included in the internet program).

Safety parameters: As a mean to monitor safety and progress participants complete two self-report measures within the program (PTSD Checklist for DSM-5 [PCL-5] and Hospital anxiety and depression scale [HADS] twice during the program and the therapist can follow these scores. In addition, participants can report any adverse events during treatment, at post treatment and follow-up assessment.

Data collection: Self-report measures will be mailed to participants

Main statistical analysis: Between-group estimates on outcome will be conducted using repeated measurements. The analyses will be conducted using intention to treat principles and post hoc comparisons.

ELIGIBILITY:
Inclusion Criteria:

* a CAPS of ≥25
* subjected to single traumatic events
* were able to understand Swedish
* had symptoms of chronic pain that interfered significantly with everyday life
* were fully examined medically and had received medical treatment if indicated
* were able to be an active part of the rehabilitation process, regain functioning in different life areas and participate in treatment interventions for approximately 5 hours every week
* stable dose of medication
* able to read and write in Swedish
* had access to a smart phone or computer with internet access

Exclusion Criteria:

* repeated and extensive traumatic events
* had other acute or severe psychiatric disorders or symptoms that warranted designation as the primary disorder (ongoing substance dependence, untreated bipolar disorder, OCD, psychotic symptoms, severe depression)
* were actively abusing analgesic medications (including narcotics), alcohol or other drugs
* had great difficulty to harbour and handle strong emotions that could lead to emotional outbursts or self-harming behavior
* had health risks due to medical reasons;
* had social or economic difficulties or lack of social support that hindered behavior change
* current severe suicidal ideation that warranted immediate intervention (indicated by the MINI and a score of 3 to item 9 of the Patient Health Questionnaire 9-item version (PHQ9))

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
PTSD diagnostic status as measured by the Clinician-Administered PTSD Scale (CAPS) | Baseline, two-week-post treatment.
  (changes between assessments) The scale assesses the presence of the DSM-5 PTSD criteria A-J.
PTSD symptom severity as measured by the the Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) and the Life Events Checklist (LEC-5) | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments) The scale ranges from 0-80 and higher sores indicate greater severity of PTSD symptoms.

SECONDARY OUTCOMES:
Anxiety and depression as measured by the Hospital Anxiety and Depression Scale (HADS) | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments) The subscales range from 0-21 and higher scores corresponds to greater severity of depression/anxiety.
Psychological inflexibility as measured by the Psychological Inflexibility in Pain Scale (PIPS) | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments) The scale ranges from 12-84 and higher scores corresponds to greater psychological inflexibility.
Acceptance as measured by the Chronic Pain Acceptance Questionnaire-8 (CPAQ-8) | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments) The scale ranges from 0-48 and higher scores corresponds to greater acceptance.
Posttraumatic Cognitions as measured by the Posttraumatic Cognitions Inventory (PTCI) | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments) The scale ranges from 33-231 and higher scores corresponds to greater endorsement of trauma-related thoughts and beliefs.
Pain interference as measured by the Multidimensional Pain Inventory (MPI) | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments) The scales ranges from 0-6 and higher scores corresponds to greater pain interference.
Pain intensity as measured by the Numerical Rating Scale (NRPS) | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments) The scale ranges from 0-10 and higher scores corresponds to greater pain intensity.
Pain catastrophizing as measured by the Pain Catastrophizing Questionnaire (PCS) | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments) The scale ranges from 0-52 and higher scores represent greater pain catastrophizing.
Perceived health as measured by the RAND-36 Measure of Health-Related Quality of Life (RAND-36) | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments) Each subscale is directly transformed into a 0-100 scale where higher scores correspond to greater levels on that specific subscale.
Kinesiophobia as measured by the Tampa Scale of Kinesiophobia (Tampa) | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments) The scale ranges from 17-68 and higher scores represent greater levels of kinesiophobia.
Number of adverse events reported by the participant | 2-week-post treatment.
Health care utilization, pharmaeconomics, medication use, and return to work as measured by the MiDAS-database of the Swedish Social Insurance Agency, the Swedish Prescribed Drug Register and health-care database of Region Skåne | Baseline, two-week-post treatment, 3 month-follow-up.
  (changes between assessments)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pain Pehabilitation, Skåne University Hospital, Lund, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akerblom S, Nilsson T, Stacke S, Peppler Jonsson I, Nordin L. Internet-based acceptance and commitment therapy for transdiagnostic treatment of comorbid posttraumatic stress disorder and chronic pain: A development pilot study. Psychol Trauma. 2025 Sep;17(6):1154-1164. doi: 10.1037/tra0001663. Epub 2024 Feb 29. PMID 38421757